CLINICAL TRIAL: NCT00460551
Title: A Randomized, Open-label, Multi-center Trial Investigating Zalutumumab, a Human Monoclonal Anti-EGF Receptor Antibody, in Combination With Chemo-Radiation in Stage IIIA-IIIB Non Small Cell Lung Cancer Patients
Brief Title: Zalutumumab in Combination With Chemo-Radiation in a Certain Type of Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to considerations regarding the appropriate therapeutic regimen for these patients.
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN204
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Results first posted 2011-12-05 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — zalutumumab; Induction Chemotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zalutumumab 8 mg/kg (Experimental)
  Interventions: Biological: Zalutumumab; Drug: Induction chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Zalutumumab — 8 mg/kg
Drug: Induction chemotherapy — Combination of cisplatin and docetaxel administered as two cycles given every three weeks
Radiation: Radiotherapy — 64 Gy in 32 fractions over 6.5 weeks

SUMMARY:
The purpose of the study is to investigate if treatment with zalutumumab in combination with chemotherapy and radiotherapy (chemo-radiation) will lead to a prolonged life in patients with lung cancer compared to patients treated with chemo-radiation alone.

DETAILED DESCRIPTION:
Originally the study was planned as Part 1A, Part 1B and Part 2. Part 1A was one arm with zalatumumab fixed dose 8 mg/kg. Part 1B was planned as zalutumumab dose-titration and Part 2 adding a comparator. The trial was prematurely closed for enrolment when patients had only been enrolled in Part 1A due to published results showing increased toxicity from induction chemotherapy without any survival benefit.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC stage IIIA-IIIB
* Performance status 0 or 1 (Zubrod or WHO Scale)

Exclusion Criteria:

* Evidence of metastases either in a separate lobe of the lung, or extra thoracic
* Patients with high risk of radiation pneumonitis and or compromised lung function
* Estimated life expectancy of less than 3 months
* Prior chemotherapy for lung cancer
* Prior radiotherapy to the chest
* Prior surgery with curative intent for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steen Lisby, MD, PHD, Study Director — Genmab employee
Locations (8):
- United States (2):
  - Towson, Maryland
  - Providence Portland Medical Center, Portland, Oregon
- Belgium (3):
  - UZ Gent, Ghent
  - CHR La Citadelle, Liège
  - CHU Sart-Tilman Domaine Universitaire du Sart-Tilman, Liège
- CHRU Reims, Hospital Maison Blanche, Reims, Cedex, France
- VU Medisch Centrum (VUMC), Amsterdam, Netherlands
- The Institute of Cancer Research and the Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zalutumumab 8 mg/kg
Started | 13
Completed | 13 (The trial was terminated after Period 1A. Only safety was measured.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age Continuous [Median (Full Range); unit: years] | 66 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  France | 2
  United States | 2
  Belgium | 6
  Netherlands | 1
  United Kingdom | 2

OUTCOME MEASURES:

1. Secondary Outcome: Adverse Events
Description: Number of participants reporting at least one adverse event
Time Frame: Up to 3 months
Population: Number of patients reporting at least one adverse event
Measure: Number; unit: participants
Arm/Group | Zalatumumab 8 mg/kg
Number analyzed (Participants) | 13
participants | 13

2. Primary Outcome: Progression Free Survival Verified by Imaging Techniques.
Description: Disease progression was planned to be confirmed using RECIST criteria J Natl Cancer Inst 2000;92:205-16
Time Frame: Until disease progression
Population: Data was not collected. Imaging scans were not taken during part 1A. The trial was prematurely closed when 13 patients were enrolled in part 1A. Scans were planned for part 1B and 2. No patients continued to part 1B and part 2.
Measure: Number; unit: Participants
Arm/Group | Zalatumumab 8 mg/kg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Zalutumumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 8 mg/kg (N=13)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 8 mg/kg (N=13)
Rash (Skin and subcutaneous tissue disorders) | 13 (241)
Constipation (Gastrointestinal disorders) | 10 (22)
Diarrhoea (Gastrointestinal disorders) | 8 (14)
Nausea (Gastrointestinal disorders) | 8 (14)
Fatigue (General disorders) | 8 (14)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (7)

LIMITATIONS AND CAVEATS:
The trial was prematurely closed. The original protocol contained Part 1A, followed by Part 1B and Part 2. The trial was terminated when 13 patients were enrolled in Part 1A. Scans for efficacy were planned for Part 1B and Part 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.